CLINICAL TRIAL: NCT03402750
Title: Heart Failure Medication Adherence Study
Brief Title: Heart Failure Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Beta Tau Chapter of Sigma Theta Tau International (Unknown)
Responsible Party: Principal Investigator, Brian McCabe, Research Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20160741
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Results first posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure
Keywords: Adherence, Medication, Prescription
MeSH Terms: conditions — Heart Failure | interventions — Electronic Prescribing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meds to Beds (Experimental): Patients receive medication in-hand at discharge from the hospital
  Interventions: Behavioral: Meds to Beds
- Standard Care (Active Comparator): Electronic prescription with patient pickup at the pharmacy
  Interventions: Behavioral: Electronic Prescription

INTERVENTIONS:
Behavioral: Meds to Beds — Medications will be delivered to patient bedside before discharge
  Arms: Meds to Beds
Behavioral: Electronic Prescription — Patient or surrogate can pick up medication from pharmacy
  Arms: Standard Care

SUMMARY:
The objective of this investigation is to pilot test a medication in-hand intervention (Meds to Beds) compared to standard care for patients with heart failure (ICD-50[all numbers]). The study will evaluate if the intervention improves adherence and physical health, and reduces hospital re-admissions. The study will provide evidence for the feasibility and acceptability of the medication-in-hand intervention.

ELIGIBILITY:
Inclusion Criteria:

* Admission diagnosis of heart failure ICD-50, including I50.1, I50.2, I50.20, I50.21, I50.22, I50.23, I50.3, I50.30, I50.31, I50.32, I50.33, I50.4, I50.40, I50.41, I50.42, I50.43, I50.8, I50.81, I50.810, I50.811, I50.812, I50.813, I50.814, I50.82, I50.83, I50.84, I50.89, I50.9, or any combination thereof
* Age 18 or older
* New York Heart Association Heart Failure Class II or Class III, with ejection fraction below 45%
* Cognitively intact, without significant psychological impairment affecting medication adherence such as dementia noted in patient record.

Exclusion Criteria:

* Medical conditions, such as active cancer or pregnancy, expected to alter heart failure medication management
* Discharged to nursing homes or hospice care, where patient may not responsible for their own adherence
* High risk of loss to follow-up, e.g., leaving the hospital against medical advice, prisoners, living in a homeless shelter, or unable to provide a phone number
* No plan to fill medications at the Jackson Memorial Hospital pharmacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian E McCabe, PhD, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meds to Beds | Standard Care
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meds to Beds | Standard Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.85 (6.54) | 58.55 (11.18) | 58.20 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 18 | 17 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 11 | 12 | 23
  Ethnicity: African American | 7 | 8 | 15
  Ethnicity: White | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Medication
Description: Adherence to medication will be reported as the number of participants that scores 12 and lower in a self-reported Adherence to Refills and Medications Scale (ARMS) Questionnaire. The questionnaire has 12 items with each item being recorded on a four-point Likert scale. The total score ranges from 12-48 with the lower score indicating better adherence.
Time Frame: Day 30
Population: 4 participants in each condition did not complete this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Meds to Beds | Standard Care
Number analyzed (Participants) | 16 | 16
Participants | 2 | 3

2. Primary Outcome: Pharmacy Refill Adherence to Medication
Description: Medication adherence will be reported as the number of participants that completed their expected pharmacy refill. Standard Care participants are expected to complete one initial fill and one refill. Meds to Beds participants are expected to complete one pharmacy refill as the initial fill is handed upon discharge.
Time Frame: Day 30
Population: Data on electronic medical record for refills of heart failure medications were only available for 10 participants in Meds to Beds and 11 in Standard Care.
Measure: Count of Participants; unit: Participants
Arm/Group | Meds to Beds | Standard Care
Number analyzed (Participants) | 10 | 11
Participants | 7 | 6

3. Secondary Outcome: Physical Health as Assessed by the Patient-Reported Outcome Measurement Information System (PROMIS) Questionnaire
Description: Physical health is measured using the 10 item PROMIS questionnaire. Responses are recorded along a 5-point Likert scale with a total score ranging from 10-50. A higher score indicates better physical health.
Time Frame: Baseline and Day 30
Population: Interviews completed at follow-up and baseline. Not all participants completed the PROMIS questionnaire at the 30-day follow up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meds to Beds | Standard Care
Number analyzed (Participants) | 20 | 20
score on a scale
  30-Day follow-up: number analyzed (Participants) | 16 | 16
  30-Day follow-up | 11.81 (4.09) | 11.50 (3.90)
  Baseline/Discharge | 8.56 (3.16) | 10.19 (3.51)

4. Secondary Outcome: Number of Participants That Received Their Medications Prior to Discharge.
Description: The program's feasibility will be evaluated by tracking whether medications can be successfully delivered (i.e., before discharge) to patients in the Meds to Beds condition. This measure will be evaluated as a proportion within the intervention condition.
Time Frame: Day 0
Population: Patients in Standard Care arm could receive delivery of medications, contrary to intentions.
Measure: Count of Participants; unit: Participants
Arm/Group | Meds to Beds | Standard Care
Number analyzed (Participants) | 20 | 20
Participants | 7 | 5

5. Secondary Outcome: Intervention Acceptance
Description: All participants will be asked one question about the acceptability of the intervention program. Responses for acceptability items will be recorded on a 10-point scale (1, very unsatisfactory - 10, very satisfactory). Dichotomized due to extreme skew. Intervention acceptance will be reported as the number of participants that provides a score of 1 and higher.
Time Frame: Day 30
Population: All participants completing follow-up interview. Not all participants completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Meds to Beds | Standard Care
Number analyzed (Participants) | 16 | 16
Participants | 10 | 9

ADVERSE EVENTS:
Time Frame: 30 days
Description: Event data collected from interview and medical records
Arm/Group | Meds to Beds | Standard Care
All-Cause Mortality (participants affected / at risk) | 1/20 | 1/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meds to Beds (N=20) | Standard Care (N=20)
Death (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03402750/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03402750/SAP_001.pdf